CLINICAL TRIAL: NCT03685006
Title: Carotid Atherosclerosis, Inflammation and Ischemic Stroke
Brief Title: Atherosclerosis and Acute Ischemic Stroke Study
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); University Hospital, Akershus (Other); Ostfold Hospital Trust (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Mona Skjelland, Consultant, Associate professor, Oslo University Hospital
Other Study IDs: REK 2009/5237
Record Dates: First submitted 2018-08-10; First posted 2018-09-26 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Atherosclerosis; Inflammation; Ischemic Stroke
MeSH Terms: conditions — Atherosclerosis; Inflammation; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Carotid artery plaques removed by carotid endartrectomy Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A significant proportion of strokes are thromboembolic in nature, arising from atherosclerotic plaque at the carotid bifurcation. It is now wellknown that inflammation plays a key role in atherogenesis and plaque destabilization. However the identification and characterization of the different inflammatory factors, as well as their relative importance, have not been clarified. This main aim of this study is to identify new risk markers for atherosclerosis and to characterize more precise methods for detection of the unstable carotid plaque with increased stroke-risk.

DETAILED DESCRIPTION:
This project include patients with asymptomatic and symptomatic carotid stenosis >50%. Patients with acute ischemic stroke will also be included with carotid artery stenosis <50% (study 3). The patient group will undergo a clinical neurological examination, ultrasound of the neck-arteries and a blood sample. The majority will also have a CT-angiography of the neck arteries and a cerebral MRI or CT. Carotid plaques removed by surgery (carotid end-arterectomy) and thrombs removed by thrombectomy will undergo histological analyses.

Study 1:

Plasma markers will be analysed and compared to clinical symptoms, ultrasound assessment of the plaque, cerebral MRI (or CT).

Study 2:

Results from advanced ultrasound of the carotid plaque including assessment of plaque morphology will be compared to histology of the removed plaque. Plasma markers and clinic will be related to the findings. The correlation between the different diagnostic modalities and the histologic conclusion will be assessed.

Study 3:

This study focus on plasma markers in an acute ischemic stroke due to a carotid plaque compared to an acute ischemic stroke with a cardial embolic source. Thrombi removed from the cerebral artery by thrombectomy will undergo histological analysis and the results will be compared to plasma markers and stroke aetiology.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an atherosclerotic carotid stenosis >50% admitting one of the study centres as an in-patient or an out-patient will be considered for inclusion.
* Acute stroke patients treated with thrombectomy at Oslo University Hospital will be included even though the carotid stenosis is < 50%.

Exclusion Criteria:

* Malign disease
* Inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with carotid atherosclerosis and/ or cerebrovascular symptoms/ disease.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Plasma markers and advanced ultrasound of neck arteries to detect plaque instability, predict stroke risk and correlation to stroke aetiology. | one year
  Blood test, ultrasound, cerebral MRI, clinical assessment

SECONDARY OUTCOMES:
Plasma markers to predict plaque instability | At inclusion
  Blood test, ultrasound, cerebral MRI
Advanced ultrasound for detection of carotid plaque instability | At inclusion and after one year
  Ultrasound, blood test, cerebral MRI, histology of carotid artery plaques
Plasma markers to determine correlation of acute ischemic stroke due to a carotid plaque compared to an acute ischemic stroke with a cardial embolic source | At inclusion
  Blood tests, ultrasound of neck arteries, cerebral MRI, histology of removed cerebral thrombi

CONTACTS AND LOCATIONS:
Overall Officials: Mona Skjelland, MD/postdoc, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway